CLINICAL TRIAL: NCT02591017
Title: Comparison of Oral Morphine Versus Nasal Ketamine Spray With Chitosan in Cancer Pain Outpatients
Acronym: ONKEMI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKNZ 2014-249
Record Dates: First submitted 2015-04-01; First posted 2015-10-29 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Cancer: Breakthrough Pain; Cancer: Extreme Pain on Movement
MeSH Terms: interventions — Morphine; Ketamine; Chitosan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- morphine drops solo and placebo spray (Other): morphine 2% drops
  1. daily fixed dose of morphine equivalents < 100 mg, 0.2 mg/kg Body weight morphine drops every hour in reserve due to international Standards
  2. daily fixed dose of morphine equivalents =/> 100 mg, 15% of the fixed daily dose in morphine drops every hour in reserve due to international standards
  Interventions: Drug: Morphine; Drug: Placebo
- ketamine/chitosan spray nasal and placebo drops (Other): 5 mg ketamine all 5 minutes, maximal 4 times an hour
  Interventions: Drug: Ketamine; Drug: Placebo; Drug: Chitosan
- morphine drops and ketamine/chitosan spray nasal (Other): see above
  Interventions: Drug: Morphine; Drug: Ketamine; Drug: Chitosan

INTERVENTIONS:
Drug: Morphine
  Arms: morphine drops and ketamine/chitosan spray nasal; morphine drops solo and placebo spray
Drug: Ketamine
  Arms: ketamine/chitosan spray nasal and placebo drops; morphine drops and ketamine/chitosan spray nasal
Drug: Placebo
  Arms: ketamine/chitosan spray nasal and placebo drops; morphine drops solo and placebo spray
Drug: Chitosan
  Arms: ketamine/chitosan spray nasal and placebo drops; morphine drops and ketamine/chitosan spray nasal

SUMMARY:
34 adult (>18 years) cancer pain outpatients with Opioid base therapy because of pain and breakthrough pain or extreme pain on movement will be included in this prospective, randomized, double-blind crossover study.

Over a period of 3 weeks patients will go through 3 treatment arms, each one lasting one week: Group A receives morphine drops and Placebo spray, Group B receives ketamine/chitosan spray nasal and Placebo drops and Group C receives morphine drops and ketamine/chitosan spray nasal.

Primary endpoint is time to onset of action of intranasal ketamine compared with morphine drops. Secondary endpoint is the median numeric rating scale (NRS) improvement after using the spray or morphine or the combination of ketamine spray and morphine drops.

ELIGIBILITY:
Inclusion Criteria:

* Cancer pain in outpatients with:
* Opioid based therapy due to pain
* Breakthrough pain or
* Extreme pain on movement
* Age >= 18 years

Exclusion Criteria:

* Patients unable to give written informed consent
* Patients unable to understand how to handle and document the use of the study medication
* Known drug allergies or intolerance to ketamine
* Known drug allergies or intolerance to morphine
* Known allergy to crustacea or chitosan
* Patients using snuff at a regular basis
* Recreational drug addiction or abuse
* Serious intranasal or epipharyngeal Problems (Septum wall defects, cancer)
* Mental/psychiatric disorder
* Patients with renal failure (clearance < 30 ml/min)
* Pregnancy and breast feeding mothers
* Patients not understanding German
* Patient having arterial hypertonia with measured values > 180/95

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02; Primary Completion 2017-07 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Time to onset of action of intranasal ketamine compared with morphine drops | 5 minutes
Time to onset of action of intranasal ketamine compared with morphine drops | 10 minutes
Time to onset of action of intranasal ketamine compared with morphine drops | 15 minutes
Time to onset of action of intranasal ketamine compared with morphine drops | 20 minutes
Time to onset of action of intranasal ketamine compared with morphine drops | 45 minutes

SECONDARY OUTCOMES:
Median NRS improvement after using the spray or morphine or the combination of ketamine spray and morphine drops | after 5, 10, 15, 20, 45 minutes
Total amount of delivered applications of ketamine or morphine in each study arm | 3 weeks
Total amount of fixed and reserve opioid doses increase in each study arm | 3 weeks
Assessment of Nausea, vomiting, itching, fatigue, hallucinations, Irritation of nasal mucosa | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wilhelm Ruppen, PD Dr. med., Principal Investigator — Pain Relief Unit and Anaesthesiology, University Hospital Basel, Switzerland
Locations (1):
- Pain Relief Unit and Anaesthesiology, University Hospital Basel, Basel, Switzerland